CLINICAL TRIAL: NCT04497610
Title: SARS-CoV-2 (COVID-19) Detection Using the Breath Analizer TeraSystem
Status: Withdrawn | Type: Observational
Why Stopped: Study was not initiated
Sponsor: Instituto Costarricense de Investigaciones Clínicas ICIC (Other)
Responsible Party: Principal Investigator, Dr. Guillermo Rodríguez Gómez, Founder, Instituto Costarricense de Investigaciones Clínicas ICIC
Other Study IDs: Tera-CR-1
Record Dates: First submitted 2020-08-02; First posted 2020-08-04 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: COVID19
Keywords: SARS-CoV-2, coronavirus testing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — breath sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive TeraSystem test: Patients having positive PCR tests will undergo TeraSystem test
  Interventions: Diagnostic Test: Breath sample
- Negative TeraSystem test: Patients having negative PCR tests will undergo TeraSystem test
  Interventions: Diagnostic Test: Breath sample

INTERVENTIONS:
Diagnostic Test: Breath sample — Patient will blow into a tube 5 times.

SUMMARY:
The purpose of the study is to verify the sensibility and accuracy of a rapid detection test for SARS-CoV-2 in breath samples analyzed by the breath detector analyzer TeraSystem, comparing with PCR tests.

DETAILED DESCRIPTION:
BioSafety Technologies has developed a rapid detection test to clear people of COVID-19.

A person can undergo an easy non-invasive test, to determine if they are: COVID-19 Clear (Negative) or Infected (Positive). The user-friendly process does not involve medically trained personnel.

The study will compare TeraSystem test results against PCR test results. Persons participating will be persons having a PCR test as part of the Health System and consenting to participate.

ELIGIBILITY:
Inclusion Criteria:

Older than 7 years odf age Able to provide informed consent Able to take the breath test

Exclusion Criteria:

Younger than 7 years of age Unable to provide informed consent Unable to take the breath test

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population under Country's screening program and known positive cases.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Presence of disease | 1 minute
  Established diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Rodríguez Gómez, MD, Principal Investigator — Founder and Investigator
Locations (1):
- Instituto Costarricense de Investigaciones Clínicas, San José, Costa Rica

IPD SHARING:
Plan to Share IPD: No
Personal data will be coded. No identifying information will be shared. Only demographic, and breath tests results will be shared.